CLINICAL TRIAL: NCT02491047
Title: Safety and Performance of BonyPid-1000™ in the Treatment of Gustilo I, II, IIIA and IIIB Tibial Open Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PolyPid Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BonyPid-1000TM-103
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Tibial Fractures; Open Fractures
MeSH Terms: conditions — Tibial Fractures; Fractures, Open | interventions — Standard of Care; Therapeutics

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into either Study investigational arm or Study control arm, using a 1:1 ratio. Randomization will be stratified by Gustilo classification (I and II; IIIA ; IIIB).
  In the study treatment arm patients will receive BonyPid-1000 in addition to the standard of care treatment. in the control arm patients will receive the standard of care treatment alone.
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- BonyPid-1000 (Experimental): Implantation of BonyPid-1000 medical device, constructed of bone filler coated with controlled release antibiotic formulation, concomitantly with standard of care treatment (SOC)
  Interventions: Device: BonyPid-1000; Other: Standard of Care (SOC) treatment
- Study control arm (Other): Standard of care treatment (SOC) only
  Interventions: Other: Standard of Care (SOC) treatment

INTERVENTIONS:
Device: BonyPid-1000 — BonyPid-1000 implantation concomitantly to standard of care (SOC) treatment
  Arms: BonyPid-1000
Other: Standard of Care (SOC) treatment — Standard of Care (SOC) treatment only

SUMMARY:
This is a prospective, multi-national, multicenter, randomized, two arms, single blind, Standard of Care (SOC) controlled, with blinded central reading center study. This study will assess the safety and performance of BonyPid-1000™ in severe open tibial fractures (Gustilo IIIA and IIIB) when implanted as adjunct to SOC and compared to SOC alone.

DETAILED DESCRIPTION:
The study population include subjects with a classification of Gustilo I, II, IIIA or IIIB of tibial open fractures, assigned for surgical procedure, who meet eligibility criteria and provide signed informed consent.

Subjects will be randomized into either Study investigational arm or Study control arm, using a 1:1 ratio. Randomization will be stratified by Gustilo classification (I and II; IIIA ; IIIB).

Total duration of the study is expected to be approximately 32 months from first subject enrolled until last subject completed.

It is expected that each subject will be in the study for approximately 52 weeks

Subjects will be followed at the following time points:

* Immediately post index procedure
* During hospitalization
* Discharge visit
* 4 weeks and then monthly up to 24 weeks, 36 and at 52 weeks.

This is a single blind clinical trial. Subjects and their family members will be blinded to the treatment arms assignment. The study site personnel present at the baseline procedure as well as the physician performing the procedure will be trained not to disclose the treatment arm to the subject, his/her family, and to health care providers outside of the Orthopedic department.

An independent X-ray reading center assessing all subjects' images will be blinded to the treatment arms assignments, for the entire trial period. However, due to the radiographic appearance of the BonyPid-1000 as compared to SOC may differ, it is not entirely possible to blind the evaluating radiologists.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female aged between 18 to 70 years of age.
2. Female of childbearing potential should have a negative urine pregnancy test prior to index procedure Note: All female of childbearing potential must agree to use a highly effective method of contraception consistently and correctly for the duration of the study.
3. Subjects with tibia open fractures of Gustilo grade I, II, IIIA or IIIB, who are assigned for surgery and are suitable for bone filler implantation, are eligible to participate in the study.
4. Single or multi-injured subjects who are hemodynamically and physiologically stable.

   Note: A multi-injured subject is defined as one who sustains ≥2 injuries, each injury requiring hospitalization, independently of the presence of other injuries.
5. Subjects who are able and willing to sign an informed consent form, prior to any protocol-specific procedures being performed and accept to comply with protocol requirements for the duration of the study. In specific cases, due to medical condition (e.g. a medical condition which necessitate an immediate medical treatment), a shortened consenting process may take place in accordance with local regulations.

Exclusion Criteria:

1. Female who is pregnant or breastfeeding.
2. Subjects with known current disseminated malignancies, active cancer or autoimmune diseases. Note: active cancer defined as - cancer for which therapeutic or palliative treatment is either ongoing at the time of enrolment or has stopped less than six (6) months before enrolment.
3. Subjects with fractures due to known medical history of Osteoporosis.
4. Subject with known medical history of Diabetes.
5. Heavy smokers (a smoker with a daily cigarettes consumption of more than 20 pieces) in the last 6 months.
6. Drug/alcohol abusers
7. Acute infection in another sites/organs.
8. Non-ambulating subjects prior to the trauma.
9. More than 24 hours between injury and systemic antibiotic treatment initiation
10. Subjects with bone fracture due to known medical history of metabolic bone diseases.
11. Subjects with high velocity gunshot bone fractures.
12. Subjects with major intra-articular fractures
13. Subjects with hypersensitivity to doxycycline and or tetracycline family of drugs.
14. Subjects treated with systemic doxycycline during the last 4 weeks prior to screening.
15. Previous surgical intervention in the target tibia
16. Subject with previous open fractures within one year in the target tibia
17. Subjects currently receiving or have received an investigational product in the last 30 days and/or participate in another clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Safety: Deep Infection in the target fracture site | During the 4 weeks post index procedure
  Deep Infection in the target fracture site during the 4 weeks post index procedure. The endpoint will be assessed by calculating the rate /percent per group.
Performance: Radiographic-assessed bone healing | During the 24-week follow-up period
  Radiographic-assessed bone healing during the 24-week follow-up period, based on independent blinded central radio-graphic evaluations of the target fracture's X-rays.

SECONDARY OUTCOMES:
Performance: Time to Radiographic-assessed bone healing | During the 24-week follow-up period
  Time to radiographic-assessed bone healing, based on independent blinded central radio-graphic evaluations of the target fracture's X-rays.

CONTACTS AND LOCATIONS:
Overall Officials: Shany Blum, Dr., Study Director — PolyPid Ltd.
Locations (9):
- Israel (6):
  - Rabin Medical Center, Petah Tikva, Central District
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital, Jerusalem
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Philippines (3):
  - De La Salle HSI, Cavite
  - Philippines General Hospital, Manila
  - Philippine Orthopedic Center, Quezon City